CLINICAL TRIAL: NCT03491618
Title: Evaluación de la Analgesia a Corto y Medio Plazo de Las Diferentes Posiciones y Tipos de Las cánulas de Radiofrecuencia, en la denervación Del Ramo Medial Del Nervio Dorsal Lumbar
Brief Title: Analgesic Effect of Different Positions and Canulae on Medial Branch Radiofrequency Denervation for Lumbar Zygapophyseal Joint Pain
Acronym: EARL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP5017
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Lumbar Facet Joint Pain; Lumbar Medial Branch Neurotomy
Keywords: lumbar facet joint pain; Lumbar Medial Branch Neurotomy; Chronic Low Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective comparative study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARALLEL (Active Comparator): Thick canulae (18 gauge) placed parallel to Medial Branch under fluoroscopy.
  Interventions: Other: PAIN REDUCTION ON VAS/NRS
- PERPENDICULAR (Active Comparator): Thin canulae (22 gauge) placed perpendicular to Medial Branch under fluoroscopy.
  Interventions: Other: PAIN REDUCTION ON VAS/NRS

INTERVENTIONS:
Other: PAIN REDUCTION ON VAS/NRS — Pain reduction comparing two different techniques and canulae placement, under fluoroscopic guidance.

SUMMARY:
Prospective study to analyse pain reduction with two types of canulae and two types of placements for lumbar medial branch radiofrequency denervation.

DETAILED DESCRIPTION:
Patients who suffer from lumbar zygapophyseal joint pain often receive radiofrequency medial branch denervation as treatment. Many types if canulae exist, and many types of placing them in relation to the Medial Branch nerves (MB). The EARL study tries to compare the analgesic effect of thin canulae (22 gauge) placed perpendicular to MB to thicker canulae (18 gauge) placed parallel to MB.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain of > 3 months
* 18-80 years
* VAS or NRS>6
* Positive controlled block

Exclusion Criteria:

* Pregnancy
* Psichiatric disorders
* Not being able to fulfil questionnaires
* Body Mass Index>35
* Labor Litigation
* Negative or non conclusive controlled block
* Failed Back Surgery Syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
PAIN REDUCTION ON VAS/NRS | 1-3-6 months
  Reduction in pain, at 1,3 and 6 months

SECONDARY OUTCOMES:
OSWESTRY DISABILITY INDEX | 1-3-6 months
  Quantify disability for low back pain.
ROLAND MORRIS | 1-3-6 months
  Health status measure for low back pain
MEDICATION REDUCTION | 1-3-6 months
  Pain medication reduction
WORKING STATUS | 1-3-6 months
  CHANGE IN WORKING STATUS

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided